CLINICAL TRIAL: NCT02212665
Title: Life Without Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Gentofte, Copenhagen (Other)
Responsible Party: Principal Investigator, Pernille Mensberg, MSc, ph.d-student, University Hospital, Gentofte, Copenhagen
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: H-4-2013-079
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Last update posted 2021-07-09 (Actual); Status verified 2021-07

CONDITIONS: Prevention of Developing Type 2 Diabetes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- High intense interval training (HIIT) (Experimental): 3 x 20 sec, 3 x week
  Interventions: Behavioral: High intense interval training
- Increased daily activity detected by the pedometer (Experimental): 10.000 steps a day
  Interventions: Behavioral: Increased daily activity detected by the pedometer
- Increased daily activity detected by te pedometer+HIIT (Experimental): 10.000 steps + 3 x 20 sec, 3 x week
  Interventions: Behavioral: Increased daily activity detected by the pedometer+HIIT
- Increased daily activity (pedometer)+group intervention (Experimental): 10.000 steps + group intervention
  Interventions: Behavioral: Increased daily activity detected by the pedometer+group intervention
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: High intense interval training
  Arms: High intense interval training (HIIT)
Behavioral: Increased daily activity detected by the pedometer
  Arms: Increased daily activity detected by the pedometer
Behavioral: Increased daily activity detected by the pedometer+HIIT
  Arms: Increased daily activity detected by te pedometer+HIIT
Behavioral: Increased daily activity detected by the pedometer+group intervention
  Arms: Increased daily activity (pedometer)+group intervention

SUMMARY:
The aim of the study 'Live - without diabetes' is to investigate the effects of increased physical activity on a daily basis with or without (high intense interval training) HIIT (short and intense: 3 minutes per week) during 12 weeks in risk individuals with pre-diabetes

DETAILED DESCRIPTION:
A total of 125 individuals with pre-diabetes will be included and randomized into four different groups (N=25, each group): 1) Increased daily activity detected by the pedometer, 2) increased daily activity detected by the pedometer + HIIT, 3) HIIT, and 4) increased daily activity detected by the pedometer + group intervention 5) a control group (maintain unchanged activity and life-style during the duration of the study).

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) > 25 kg/m2
* Prediabetes: 6.1 % ≤ glycated hemoglobin A1c (HbA1c) ≤ 6.4 % and / or increased fasting plasma glucose (FPG): 6.1 mM ≤ FPG ≤ 6.9 mM and / or abnormal glucose tolerance (7.8 mM ≤ 2 hour plasma glucose (PG) ≤ 11.0 mmol)
* Weekly training status <150 minutes

Exclusion Criteria:

* BMI <25 kg/m2
* Diabetes
* Pregnancy and breastfeeding
* Treatment with medicine, there influence glucose metabolism
* Decreased liver function (liver transaminases > 3 times of limit of normal)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2014-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Changes in insulin sensitivity | At baseline and after 12 weeks
  The primary endpoint is insulin sensitivity, and it will be assessed by changes in the area under the curve from baseline to end-of-study assessed by the Cederholm Index and Matsuda Index

SECONDARY OUTCOMES:
Changes in oxygen peak oxygen uptake | At baseline and after 12 weeks
  Assessed from a physical fitness test (VO2peak)
Changes in glycaemic control | At baseline and after 12 weeks
  Measured as fasting plasma glucose, HbA1c
Changes in key proteins in glucose and fat metabolism (Skeletal muscle) | At baseline and after 12 weeks
  Expression/content of key proteins in skeletal muscle tissure (AU units)
Changes in body weight (kg) | At baseline and after 12 weeks
  Measured by Dual-energy X-ray Absorptiometry, DXA
Changes in key proteins in glucose and fat metabolism (Adipose fat tissure) | At baseline and after 12 weeks
  Expression/content of key proteins in adipose tissue (AU units)
Patient-reported outcome measure | At baseline and after 12 weeks
  Health related quality of life measured from Short Form 36 (SF36). Where scores are presented as norm-based scores (0-100) with higher scores indicating better perceived health status.

CONTACTS AND LOCATIONS:
Locations (1):
- Center for Diabetes Research, Gentofte Hospital, Hellerup, Denmark